CLINICAL TRIAL: NCT05605743
Title: Ocular Hypertension Response to Alternate Nostril Breathing Training in Geriatrics With Glaucoma and High Blood Pressure
Brief Title: Alternate Nostril Breathing Training in Geriatrics With Glaucoma and High Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004006
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Primary Open Angle Glaucoma; Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Hypertension | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): Thirty hypertensive geriatric with high tension type primary open angle glaucoma will perform breathing exercise (alternate nostril breathing). The daily breathing exercise will be performed by the geriatrics in evening (for half an hour) and morning (for half an hour) for one month.
  Interventions: Behavioral: breathing exercise
- control group (No Intervention): this will be a thirty-patient wait-list group that will no receive any shape of training

INTERVENTIONS:
Behavioral: breathing exercise — Thirty hypertensive geriatric with high tension type primary open angle glaucoma will perform breathing exercise (alternate nostril breathing). The daily breathing exercise will be performed by the geriatrics in evening (for half an hour) and morning (for half an hour) for one month.
  Arms: Exercised group

SUMMARY:
Hypertension, particularly if poorly controlled, appears related to an increased risk of open angle glaucoma, (the high tension type of glaucoma is characterized as optic nerve degeneration with ocular hypertension). so this study will search response of glaucoma to breathing exercise

DETAILED DESCRIPTION:
Hypertension, particularly if poorly controlled, appears related to an increased risk of open angle glaucoma, (the high tension type of glaucoma is characterized as optic nerve degeneration with ocular hypertension). With a random assignment, sixty hypertensive geriatric with high tension type primary open angle glaucoma will be assigned to breathing exercise (alternate nostril breathing) group (n=30 geriatrics) or waiting list geriatrics. the daily breathing exercise will be performed by the geriatrics in evening (for half an hour) and morning (for half an hour).

ELIGIBILITY:
Inclusion Criteria:

* hypertensive elderly
* primary open angle glaucoma in both eyes
* ocular hypertension in both eyes

Exclusion Criteria:

acute or chronic eye inflammation cataract eye surgeries mental ill patients patients who will refuse to participate in the study other systemic /cardiovascular problem

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
intraoccular pressure | It will be measured after 4 weeks of training
  it will be measured in right and left eyes

SECONDARY OUTCOMES:
systolic blood pressure | It will be measured after 4 weeks of training
  it will be measured sphygmomanometer
diastolic blood pressure | It will be measured after 4 weeks of training
  it will be measured sphygmomanometer
heart rate | It will be measured after 4 weeks of training
  it will be measured manually
respiratory rate | It will be measured after 4 weeks of training
  it will be measured manually
hospital anxiety and depression scale | It will be measured after 4 weeks of training
  it contains fourteen questions. it contains two sub-scales, one for anxiety and the other for depression
short form 36 survey | It will be measured after 4 weeks of training
  in general, it will assess life quality
glaucoma quality of life-15 questionnaire | It will be measured after 4 weeks of training
  it will assess glaucoma-related life quality

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt